CLINICAL TRIAL: NCT03428334
Title: A 4-week Single-arm Study of Roflumilast in Stable-state Non-cystic Fibrosis Bronchiectasis
Brief Title: Roflumilast in Non-CF Bronchiectasis Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Chung-Man HO, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROF2017_v1
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: Sputum leukocyte density
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral roflumilast (Experimental): oral roflumilast 500 microgram daily for 4 weeks
  Interventions: Drug: Oral roflumilast

INTERVENTIONS:
Drug: Oral roflumilast — Roflumilast, a phosphodiesterase 4 (PDE4) inhibitor is approved worldwide (including Hong Kong) for treatment of severe chronic obstructive pulmonary disease (COPD) with frequent exacerbations. Roflumilast has been shown to have anti-inflammatory effect in patients with COPD, with significant reduction of sputum absolute neutrophil count, IL-8 and neutrophil elastase compared with placebo treatment. Roflumilast can also improve the lung function parameters in patients with COPD and reduce the rate of moderate-to-severe exacerbations.
  Other Names: Daxas

SUMMARY:
This is a single-arm, open label, Phase II study of Roflumilast in stable-state non-cystic fibrosis bronchiectasis subjects.

Bronchiectasis refers to a suppurative lung condition characterized by pathological dilatation of bronchi. The predominant aetiology of bronchiectasis in the Western population is related to cystic fibrosis (CF), which is genetically determined. Bronchiectasis due to other causes are generally grouped under the term "non-CF bronchiectasis", which accounts for practically all cases that are seen commonly in Hong Kong and many other Chinese populations.

The main pathogenesis of non-CF bronchiectasis involves airway inflammation, abnormal mucus clearance and bacterial colonization, resulting in progressive airway destruction and distortion. The current treatment strategies mainly focus on targeting the key elements in the pathogenesis of non-CF bronchiectasis.

In patients with bronchiectasis, there is also neutrophilic inflammation as in COPD. It is hypothesized that roflumilast can improve airway inflammation, sputum volume and sputum inflammatory markers in patients with bronchiectasis.

This study aims to investigate the effect of short-term (4-week) treatment with roflumilast on neutrophilic airway inflammation in stable-state non-CF bronchiectasis.

DETAILED DESCRIPTION:
Apart from regular chest physiotherapy and postural drainage to help clearing mucus from bronchiectatic airways, inhalational and parenteral antibiotics have also been used to reduce the bacterial load in destroyed airways, thus controlling and preventing infective exacerbations. In recent years, accumulated evidence has suggested a central role of airway inflammation and immune dysregulation in the evolution of non-CF bronchiectasis. The classical type of airway inflammation is neutrophilic, with abundance of neutrophils in sputum, bronchoalveolar lavage fluid and bronchial biopsy from patients with non-CF bronchiectasis, even in clinically stable-state. The recruitment and trafficking of neutrophils to bronchiectatic airways are mediated via various pro-inflammatory cytokines like interleukin-1β (IL-1β), IL-8, tumour necrosis factor (TNF)-alpha and leukotriene B4 (LTB4). Investigators have also shown in an in vitro model that sputum from patients with non-CF bronchiectasis could stimulate IL-6 production from normal human bronchial epithelial cells, mediated via TNF-alpha. Recent data have suggested the involvement of Th17 immunity, in which Th17-polarized Cluster of Differentiation 4 (CD4) T cells can respond to bacteria (especially Pseudomonas aeruginosa) in bronchiectatic airways by elaboration of IL-17, leading to downstream IL-8 release from airway epithelial cells, neutrophil chemotaxis, mucus hypersecretion and formation of ectopic lymphoid follicles. This IL-17 driven pathway can further aggravate the vicious circle of key pathogenetic mechanisms in non-CF bronchiectasis. In previous studies, airway neutrophilic inflammation as indicated by sputum neutrophil count was inversely correlated with lung function (forced expiratory volume in 1 second, FEV1) and directly with duration of disease and severity (Bronchiectasis Severity Score, BSI) in stable non-CF bronchiectasis. Investigators have also demonstrated that sputum elastase, released from airway neutrophils, significantly correlated with 24-hour sputum volume, number of bronchiectatic lobes, percent predicted FEV1, and sputum leukocyte count in stable-state bronchiectasis. Patients with non-CF bronchiectasis harbouring Pseudomonas aeruginosa showed greater sputum neutrophilia and volume, with lower FEV1 and FEV1/forced vital capacity (FVC) ratio in previous studies from our group and others.

This study aims to investigate the extent of airway inflammation in non-CF bronchiectasis is indicated by sputum leukocyte density (primary outcome measure), pro-inflammatory cytokines (IL-1β, IL-8, TNF-alpha, LTB4 and IL-17) and neutrophil elastase. Investigators hypothesize that 4-week treatment of roflumilast in stable-state non-CF bronchiectasis can result in: (1) reduction in sputum leukocyte density (primary hypothesis); (2) reduction in sputum pro-inflammatory cytokines (IL-1β, IL-8, TNF-alpha, and IL-17) and LTB4; (3) reduction in sputum neutrophil elastase; (4) reduction in 24-h sputum volume; (5) no change in sputum bacterial colonization, load and microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above, male or female.
2. Never-smokers or those who have smoked less than 100 cigarettes in their lifetime.
3. Confirmed diagnosis of non-CF bronchiectasis based on high-resolution computed tomography (HRCT) scan.
4. Significant sputum production (≥ 10 ml per day).
5. In stable-state bronchiectasis with no change in regular medications (e.g. inhaled steroid, macrolide) or exacerbations in the past 3 months.
6. Written informed consent obtained.

Exclusion Criteria:

1. Eversmokers (≥ 100 cigarettes in their lifetime).
2. Known chronic obstructive pulmonary disease or asthma.
3. Moderate to severe liver impairment (Child-Pugh B or C).
4. Known psychiatric illness with increased suicidal risks.
5. Body-mass index below 20 kg/m2.
6. Concomitant use of strong cytochrome P450 inducers (e.g. rifampicin, phenobarbital, carbamazepine, phenytoin).
7. Patients who are hypersensitive to roflumilast or its constituents.
8. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
sputum leukocyte density | Reduction of sputum leukocyte density in 4 weeks
  Sputum leukocyte density is measured within 2 hours of collection by a designated technician, based on five aliquots chosen randomly from the center of a fresh specimen, which are then serially diluted with phosphate-buffered saline (PBS) and read with a light microscope and a hemocytometer

CONTACTS AND LOCATIONS:
Overall Officials: James CM Ho, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong